CLINICAL TRIAL: NCT00970216
Title: A Prospective, Observational, Single-center Post-marketing Surveillance Study of Telbivudine in Chronic Hepatitis B Adults With HBeAg Positive/Negative.
Brief Title: Study of Telbivudine in Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMST-Y-1
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis B
Keywords: HBV DNA non-detectability
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be stored at screening/baseline and complete study after corresponding with inclusion/exclusion criteria.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Telbivudine — Post-marketing observation for chronic hepatitis B patients receiving Telbivudine treatment
  Other Names: Sebivo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and antiviral efficacy of telbivudine by maintained suppression of hepatitis B virus (HBV) DNA (<=300 copies/ml or 60IU/ml, undetectable by current polymerase chain reaction (PCR) - based assays) in HBeAg positive/negative patients at physician's general practice.

DETAILED DESCRIPTION:
Primary objective: To evaluate the antiviral efficacy of telbivudine by maintained suppression of HBV DNA(<=300 copies/ml or 60 IU/ml,undetectable by current PCR-based assays) in HBeAg positive patients from Week 24 to Week 48.

Methodology: This will be an open-label, prospective, observational, single-center and single arm post marketing surveillance study.

Number of patients: It is estimated to enroll 240 intent-to-treat patients in Taiwan.

Population: Male or female patients, at least 18 years of age diagnosed with chronic hepatitis B with liver disease and telbivudine is prescribed by physicians based on clinical justification. And patients are able to communicate well, provide written informed consent, and willing to participate in the entire study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age.
2. Documented chronic hepatitis B defined by all of the following:

   * Clinical history compatible with chronic hepatitis B.
   * Detectable serum hepatitis B surface antigen >= 6 months at screening visit, with either HBeAg positive or negative.
3. Willing and able to comply with the observational drug regimen and all other study requirements.
4. Willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

1. Females who are pregnant,intending to become pregnant or breast feeding.
2. Patients with co-infection with hepatitis C virus, hepatitis D virus or human immunodeficiency virus.
3. Patients with hypersensitivity to telbivudine or to any of the excipients.
4. One or more known primary or secondary causes of liver disease other than hepatitis B (e.g., alcoholism, steatohepatitis, autoimmune hepatitis, hemochromatosis, alpha-1 anti-trypsin deficiency, Wilson's disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease). Gilbert's syndrome and Dubin-Johnson syndrome will not exclude patients from participation in this trial.
5. Enrolled or planning to be enrolled in another clinical trial of an investigational agent while participating in this study.
6. Unable to receive safety and tolerability assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients, at least 18 years of age diagnosed with chronic hepatitis B with liver disease and telbivudine is prescribed by physicians based on clinical justification. And patients are able to communicate well, provide written informed consent, and willing to participate in the entire study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2009-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chau-ting Yeh, MD,PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, LinKou, Taoyuan County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin CL, Chien RN, Yeh C, Hsu CW, Chang ML, Chen YC, Yeh CT. Significant renoprotective effect of telbivudine during preemptive antiviral therapy in advanced liver cancer patients receiving cisplatin-based chemotherapy: a case-control study. Scand J Gastroenterol. 2014 Dec;49(12):1456-64. doi: 10.3109/00365521.2014.962604. Epub 2014 Oct 6. PMID 25283499

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Hepatitis B: Patients with chronic hepatitis B, who received Telbivudine treatment
Period: Overall Study
Arm/Group | Chronic Hepatitis B
Started | 160
Completed | 80
Not Completed | 80

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Hepatitis B
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 150
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 131
Region of Enrollment [Number; unit: participants]
  Taiwan | 160

OUTCOME MEASURES:

1. Primary Outcome: HBV-DNA < 300 Copies/mL in 48 Weeks
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Chronic Hepatitis B
Number analyzed (Participants) | 160
participants | 79

ADVERSE EVENTS:
Arm/Group | Chronic Hepatitis B
Serious Adverse Events (participants affected / at risk) | 0/160
Other Adverse Events (participants affected / at risk) | 78/160
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Hepatitis B (N=160)
Fever, mild (General disorders) | 5 (5)
Muscle skeleton discomfort (Musculoskeletal and connective tissue disorders) | 18 (29)
Skin rash and itching (Skin and subcutaneous tissue disorders) | 5 (6)
Dizziness and headache (Nervous system disorders) | 12 (26)
Abdominal discomfort (Gastrointestinal disorders) | 19 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Palpitation (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No